CLINICAL TRIAL: NCT06202560
Title: Effectiveness and Safety of Tofacitinib in Patients With Recalcitrant Frontal Fibrosing Alopecia : A Pilot Study
Acronym: Tofacitinib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dermatology, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/IEC 022/2566
Record Dates: First submitted 2023-11-26; First posted 2024-01-11 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Frontal Fibrosing Alopecia; Lichen Planopilaris of Scalp
Keywords: Tofacitinib; Frontal Fibrosing Alopecia Severity Index (FFASI); Frontal Fibrosing Alopecia Severity Score (FFASS); Lichen Planopilaris Activity Index (LPPAI); Frontal fibrosing alopecia; Lichen planopilaris
MeSH Terms: conditions — Lichen Planus | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofacitinib (Experimental): taking oral Tofacitinib 5 mg twice a day for 12 weeks
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — Participants in the research will receive oral Tofacitinib medication with a dosage of 5 mg, twice a day, for 12 weeks. They will be scheduled to come for follow-up every 4 weeks throughout the 12-week period, and will continue to be followed up for 4 weeks after stopping the medication. The total duration of the research will be 16 weeks. The purpose is to evaluate the effectiveness and safety of the medication.
  Other Names: Xeljanz

SUMMARY:
This study aims to determine the efficacy and safety of tofacitinib therapy in Thai patients with recalcitrant frontal fibrosing alopecia.

The main questions are

1. Does Tofacitinib significantly reduce Frontal Fibrosing Alopecia Severity Index (FFASI), Frontal Fibrosing Alopecia Severity Score (FFASS), Lichen Planopillaris Activity Index (LPPAI) compared to baseline and after 16 weeks?
2. Is Tofacitinib significantly different for adverse events compared to baseline and after 16 weeks? Participants will have a check-up in clinical and investigation and then get prescribed oral Tofacitinib 5 mg twice a day for 12 weeks. After that, they will have follow-up every 4 weeks until week 16.

DETAILED DESCRIPTION:
1.The researcher collects personal data, including age, gender, weight, height, body mass index, waist circumference, personal medical history, history of medication use in the past 3 months (menstruation history for female subjects), and records of symptoms such as hair loss history and diagnosis, pattern of hair loss on the scalp or other areas, comorbidities, family history, and other accompanying symptoms.

2. The researchers require the patients to undergo various blood tests before treatment.

3. The researchers collect data on the patients' skin conditions using a Digital Camera and a Dermoscope. They capture images of the scalp, eyebrows, eyelashes, facial rashes, joint folds, arms, legs, nails, mouth, and dark spots (if present).

4. Participants in the research will receive oral Tofacitinib medication with a dosage of 5 mg twice a day for 12 weeks. They will be scheduled to come for follow-up every 4 weeks throughout the 12 weeks, and will continue to be followed up for 4 weeks after stopping the medication. The total duration of the research will be 16 weeks. The purpose is to evaluate the effectiveness and safety of the medication.

1. The disease symptoms to be assessed include facial papule, LP pigmentosus, pruritus, trichodynia, perifollicular erythema, and hyperkeratosis.
2. Frontal Fibrosing Alopecia Severity Index (FFASI)
3. Frontal Fibrosing Alopecia Severity Score (FFASS)
4. Lichen Planopillaris Activity Index (LPPAI)
5. The photograph will be taken. The areas photographed include the scalp, eyebrows, eyelashes, facial rashes, joint folds, arms, legs, nails, dark spots (if present), and mouth. Two expert physicians will evaluate the photographs independently. The photographs of 10 patients were assessed to determine the consistency among the physicians before evaluating the actual patients. The evaluation will determine whether the patient's conditions have improved, remained stable, or worsened.
6. Dermoscopy will be performed. The areas examined include the scalp, eyebrows, eyelashes, facial rashes, joint folds, arms, legs, nails, dark spots (if present), and mouth.
7. The patient's abnormal symptoms after medication administration will be evaluated, including respiratory tract infections, skin abnormalities, gastrointestinal abnormalities, urinary tract infections, or other symptoms.
8. Laboratory tests will be conducted at weeks 4, 12, and 16 to assess the medication's safety.

ELIGIBILITY:
Inclusion Criteria:

1. Thai males or females who were at least 18 years old
2. Participants who were diagnosed with frontal fibrosing alopecia The criteria for the diagnosis of frontal fibrosis alopecia are 2 major criteria or 1 major criterion plus 2 minor criteria. (Vañó-Galván et al., 2014)
3. Participants who were diagnosed with recalcitrant frontal fibrosing alopecia

   * The patient who fails treatment of at least one drug, such as hydroxychloroquine, and/or receives others, such as immunosuppressive drugs, pioglitazone, and retinoids. However, the symptoms of FFA still appear, such as perifollicular erythematous and/or scale, after taking treatment for more than 3 months
   * The patient continued taking the medicine as prescribed and coming to follow-up
   * The patient still has the medical record, such as a picture and dermoscopy
   * The patient does not need a washout time from the current medicine

Exclusion Criteria:

1. Patients who were diagnosed with a disease that may relate to hair growth within six months, such as thyroid disease, iron deficiency anemia, liver disease, heart disease, neurological system disease, gastroenteritis disease, sexual disease, cancer, and psychologic disease
2. Pregnancy
3. Patients who have contraindications to take oral Tofacitinib such as severe infection, allergy to Tofacitinib, venous thromboembolism, leukopenia, severe liver disease, severe kidney failure, pneumonia, cancer
4. Patients who received strong or moderate to strong CYP3A4 agents
5. Patients who had positive on HBsAg and/or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chinmanat Lekhavat, MD, Study Director — Institute of Dermatology
Locations (1):
- Hair and Nail center, Institute of Dermatology, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Autrup H, Thurlow BJ, Warwick GP. The effects of the continuous administration of N,N-dimethyl-4-phenylazoaniline (DAB) on the activities and the inducibilities of some drug-metabolizing enzymes in rat liver. Chem Biol Interact. 1975 Nov;11(5):313-28. doi: 10.1016/0009-2797(75)90001-0. PMID 148
- [Background] Alves de Medeiros AK, Speeckaert R, Desmet E, Van Gele M, De Schepper S, Lambert J. JAK3 as an Emerging Target for Topical Treatment of Inflammatory Skin Diseases. PLoS One. 2016 Oct 6;11(10):e0164080. doi: 10.1371/journal.pone.0164080. eCollection 2016. PMID 27711196
- [Background] Banka N, Mubki T, Bunagan MJ, McElwee K, Shapiro J. Frontal fibrosing alopecia: a retrospective clinical review of 62 patients with treatment outcome and long-term follow-up. Int J Dermatol. 2014 Nov;53(11):1324-30. doi: 10.1111/ijd.12479. Epub 2014 Apr 16. PMID 24738979
- [Background] Binnion PF, Das Gupta R. Prophylactic antiarrhythmic drug therapy in acute myocardial infarction. Cardiovasc Clin. 1975;7(2):203-17. No abstract available. PMID 145
- [Background] Childs JM, Sperling LC. Histopathology of scarring and nonscarring hair loss. Dermatol Clin. 2013 Jan;31(1):43-56. doi: 10.1016/j.det.2012.08.001. Epub 2012 Sep 26. PMID 23159175
- [Background] Chern CJ, Beutler E. Biochemical and electrophoretic studies of erythrocyte pyridoxine kinase in white and black Americans. Am J Hum Genet. 1976 Jan;28(1):9-17. PMID 2009
- [Background] Craiglow BG, King BA. Tofacitinib Citrate for the Treatment of Vitiligo: A Pathogenesis-Directed Therapy. JAMA Dermatol. 2015 Oct;151(10):1110-2. doi: 10.1001/jamadermatol.2015.1520. PMID 26107994
- [Background] Ehrhart IC, Parker PE, Weidner WJ, Dabney JM, Scott JB, Haddy FJ. Coronary vascular and myocardial responses to carotid body stimulation in the dog. Am J Physiol. 1975 Sep;229(3):754-60. doi: 10.1152/ajplegacy.1975.229.3.754. PMID 2017
- [Background] Gupta AK, Daigle D, Abramovits W, Vincent KD. XELJANZ (Tofacitinib) for Chronic Plaque Psoriasis. Skinmed. 2015 May-Jun;13(3):227-9. No abstract available. PMID 26380510
- [Background] Harries MJ, Meyer K, Chaudhry I, E Kloepper J, Poblet E, Griffiths CE, Paus R. Lichen planopilaris is characterized by immune privilege collapse of the hair follicle's epithelial stem cell niche. J Pathol. 2013 Oct;231(2):236-47. doi: 10.1002/path.4233. PMID 23788005
- [Background] Hashmi AA, Rashid K, Ali R, Dowlah TU, Ali AH, Diwan MA, Malik UA, Irfan M, Zia S, Ahmad A. Clinicopathological Features of Alopecia With an Emphasis on Etiology and Histopathological Characteristics of Scarring Alopecia. Cureus. 2022 Aug 3;14(8):e27661. doi: 10.7759/cureus.27661. eCollection 2022 Aug. PMID 36072194
- [Background] Ho A, Shapiro J. Medical therapy for frontal fibrosing alopecia: A review and clinical approach. J Am Acad Dermatol. 2019 Aug;81(2):568-580. doi: 10.1016/j.jaad.2019.03.079. Epub 2019 Apr 3. PMID 30953702
- [Background] Ibrahim O, Bayart CB, Hogan S, Piliang M, Bergfeld WF. Treatment of Alopecia Areata With Tofacitinib. JAMA Dermatol. 2017 Jun 1;153(6):600-602. doi: 10.1001/jamadermatol.2017.0001. PMID 28355451
- [Background] Kerkemeyer KLS, Eisman S, Bhoyrul B, Pinczewski J, Sinclair RD. Frontal fibrosing alopecia. Clin Dermatol. 2021 Mar-Apr;39(2):183-193. doi: 10.1016/j.clindermatol.2020.10.007. Epub 2020 Oct 17. PMID 34272007
- [Background] Kossard S. Postmenopausal frontal fibrosing alopecia. Scarring alopecia in a pattern distribution. Arch Dermatol. 1994 Jun;130(6):770-4. PMID 8002649
- [Background] Syed HA, Idoudi S. Frontal Fibrosing Alopecia. 2024 Jun 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519001/ PMID 30085543
- [Background] Liu LY, King BA. Tofacitinib for the Treatment of Severe Alopecia Areata in Adults and Adolescents. J Investig Dermatol Symp Proc. 2018 Jan;19(1):S18-S20. doi: 10.1016/j.jisp.2017.10.003. PMID 29273099
- [Background] MacDonald A, Clark C, Holmes S. Frontal fibrosing alopecia: a review of 60 cases. J Am Acad Dermatol. 2012 Nov;67(5):955-61. doi: 10.1016/j.jaad.2011.12.038. Epub 2012 Apr 13. PMID 22503342
- [Background] Yang CC, Khanna T, Sallee B, Christiano AM, Bordone LA. Tofacitinib for the treatment of lichen planopilaris: A case series. Dermatol Ther. 2018 Nov;31(6):e12656. doi: 10.1111/dth.12656. Epub 2018 Sep 27. PMID 30264512
- [Background] Mamolo C, Harness J, Tan H, Menter A. Tofacitinib (CP-690,550), an oral Janus kinase inhibitor, improves patient-reported outcomes in a phase 2b, randomized, double-blind, placebo-controlled study in patients with moderate-to-severe psoriasis. J Eur Acad Dermatol Venereol. 2014 Feb;28(2):192-203. doi: 10.1111/jdv.12081. Epub 2013 Jan 7. PMID 23294276
- [Background] Papp KA, Menter A, Strober B, Langley RG, Buonanno M, Wolk R, Gupta P, Krishnaswami S, Tan H, Harness JA. Efficacy and safety of tofacitinib, an oral Janus kinase inhibitor, in the treatment of psoriasis: a Phase 2b randomized placebo-controlled dose-ranging study. Br J Dermatol. 2012 Sep;167(3):668-77. doi: 10.1111/j.1365-2133.2012.11168.x. PMID 22924949
- [Background] Rakowska A, Gradzinska A, Olszewska M, Rudnicka L. Efficacy of Isotretinoin and Acitretin in Treatment of Frontal Fibrosing Alopecia: Retrospective Analysis of 54 Cases. J Drugs Dermatol. 2017 Oct 1;16(10):988-992. PMID 29036252
- [Background] Sperling LC, Cowper SE. The histopathology of primary cicatricial alopecia. Semin Cutan Med Surg. 2006 Mar;25(1):41-50. doi: 10.1016/j.sder.2006.01.006. PMID 16616302
- [Background] Szymonowicz M, Lowkis B. In vitro testing method of polymers candidate destined for contact with blood. Polim Med. 1990;20(1-4):43-55. PMID 2151779
- [Background] To D, Beecker J. Frontal Fibrosing Alopecia: Update and Review of Challenges and Successes. J Cutan Med Surg. 2018 Mar/Apr;22(2):182-189. doi: 10.1177/1203475417736279. Epub 2017 Oct 23. PMID 29056083
- [Background] Van Gorkom HJ, Pulles MP, Wessels JS. Light-induced changes of absorbance and electron spin resonance in small photosystem II particles. Biochim Biophys Acta. 1975 Dec 11;408(3):331-9. doi: 10.1016/0005-2728(75)90134-6. PMID 62
- [Background] Vano-Galvan S, Molina-Ruiz AM, Serrano-Falcon C, Arias-Santiago S, Rodrigues-Barata AR, Garnacho-Saucedo G, Martorell-Calatayud A, Fernandez-Crehuet P, Grimalt R, Aranegui B, Grillo E, Diaz-Ley B, Salido R, Perez-Gala S, Serrano S, Moreno JC, Jaen P, Camacho FM. Frontal fibrosing alopecia: a multicenter review of 355 patients. J Am Acad Dermatol. 2014 Apr;70(4):670-678. doi: 10.1016/j.jaad.2013.12.003. Epub 2014 Feb 5. PMID 24508293
- [Background] Xing L, Dai Z, Jabbari A, Cerise JE, Higgins CA, Gong W, de Jong A, Harel S, DeStefano GM, Rothman L, Singh P, Petukhova L, Mackay-Wiggan J, Christiano AM, Clynes R. Alopecia areata is driven by cytotoxic T lymphocytes and is reversed by JAK inhibition. Nat Med. 2014 Sep;20(9):1043-9. doi: 10.1038/nm.3645. Epub 2014 Aug 17. PMID 25129481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recalcitrant frontal fibrosing alopecia patients who were confirmed diagnosed. Participants were out-patients treated at the Hair and Nail Center, the Institute of Dermatology, from November 2023 to March 2024 and qualified for inclusion criteria.
Pre-assignment Details: If abnormal blood test results are found during each follow-up visit, such as a 3-fold increase in liver enzymes (AST and/or ALT) from the baseline, consideration should be given to stop taking tofacitinib immediately.
Groups:
- Tofacitinib: oral tofacitinib 5 mg twice a day for 12 weeks
  Participants in the research will receive oral Tofacitinib medication with a dosage of 5 mg twice a day for 12 weeks. They will be scheduled to come for follow-up every 4 weeks throughout the 12 weeks and will continue to be followed up for 4 weeks after stopping the medication. The total duration of the research will be 16 weeks. The purpose is to evaluate the effectiveness and safety of the medication.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tofacitinib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  asian | 11
Region of Enrollment [Number; unit: participants]
  Thailand | 11

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Oral Tofacitinib in Recalcitrant Frontal Fibrosing Alopecia(FFA)
Description: The effectiveness of this study will be evaluated by comparing the Frontal Fibrosing Alopecia Severity Index (FFASI) (Max score = 100 and Min score = 0), Frontal Fibrosing Alopecia Severity Score (FFASS) (Max score = 25 and Min score = 0), and Lichen Planopilaris Activity Index (LPPAI) (Max score = 10 and Min score = 0) between week 0 (baseline week) and week 16. If a patient has a lower score on all of these indices, it means the treatment is more effective. In addition, two expert physicians will independently evaluate the photographs. The two evaluators will determine whether the patient's conditions have improved, remained stable, or worsened.
Time Frame: 16 weeks after taking oral Tofacitinib
Population: The effectiveness of tofacitinib for FFA was assessed by comparing the Frontal Fibrosing Alopecia Severity Index (FFASI) (ranging from 0 to 100), Frontal Fibrosing Alopecia Severity Score (FFASS) (ranging from 0 to 25), and Lichen Planopilaris Activity Index (LPPAI) (ranging from 0 to 10) between baseline (week 0) and week 16. Lower scores across these indices indicated greater treatment effectiveness. Two independent dermatologists reviewed patient photographs to determine improvements.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 11
score on a scale
  FFASI at baseline (week 0) | 47.5 (13.25)
  FFASI at week 16 | 44 (13.5)
  FFASS at baseline (week 0) | 16.3 (4.07)
  FFASS at week 16 | 15.9 (4.62)
  LPPAI at baseline (week 0) | 1.83 (1.01)
  LPPAI at week 16 | 1.33 (0.49)

2. Secondary Outcome: Clinical & Investigation Safety of Oral Tofacitinib in Recalcitrant (FFA)
Time Frame: 16 weeks after taking oral Tofacitinib
Measure: Number; unit: participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 11
participants
  mild acne vulgaris | 4
  hypercholesterolemia | 5

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (N=11)
hypercholesterolemia (Investigations) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 4 (5)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatique (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT06202560/Prot_SAP_000.pdf